CLINICAL TRIAL: NCT03293888
Title: Pilot Study Utilizing a Spectral Analysis Probe to Identify Glioblastoma Cells in Patients With Glioblastoma Undergoing Standard Surgical Resection
Brief Title: Spectral Analysis Probe to Identify Glioblastoma Cells
Status: Terminated | Type: Observational
Why Stopped: PI Relocation
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Other Study IDs: 8285
Record Dates: First submitted 2017-09-12; First posted 2017-09-26 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Glioblastoma
Keywords: Spectral Diagnosis Probe; Chaos Wand; Spectral Analysis; Optical Spectroscopy
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue from surgically resected tumor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a pilot, observational study to evaluate the intraoperative sensitivity of the Chaos Wand in detecting tumor tissue with glioblastoma disease.

DETAILED DESCRIPTION:
This is a pilot study to investigate if the Chaos Wand Spectral Diagnosis Probe can be used to identify Glioblastoma (GBM) cancer cells in patients undergoing standard surgical resection. Eligible patients who have consented to the use of the Chaos Wand will be scheduled for surgery as standard cancer care for GBM. During the surgical procedure, the Chaos Wand Spectral Diagnosis Probe will be utilized. Fifteen intraoperative readings and signal recordings of GBM tissue will be taken. The wand will only be used in areas that have already been deemed in need of resection due to GBM disease. Each site identified for spectral analysis will be marked. The wand does not come into contact with the brain at any point during this procedure. Following surgical resection of the GBM tumor, tissue will be collected from the same 15 sites where the Chaos Wand was used. The pathology report will be compared with the results of spectral analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female and over 18 years of age.
2. Patients with histologically proven GBM who are newly diagnosed and eligible to undergo surgical treatment or patients who are suspected of having glioblastoma on pre-operative imaging which is subsequently confirmed by histopathology following tumor resection.
3. Patients must be able to understand and willing to sign the informed consent document.

Exclusion Criteria:

1. Patients with absence of glioblastoma.
2. Patients who are not undergoing tumor resection.
3. Patients who have prior brain radiotherapy
4. Patients who have prior systemic chemotherapy
5. Patients who are not willing to sign the informed consent and agree to participate.
6. Patients who are pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes adult patients from the outpatient neurosurgery clinic or those who have presented through the University of Oklahoma emergency department and have been diagnosed with glioblastoma or are suspected of having glioblastoma based on pre-operative imaging. The Stephenson Cancer Center will not exclude potential subjects from participating in this or any study solely on the basis of ethnic origin or socioeconomic status. Every attempt will be made to enter all eligible patients into this protocol and therefore address the study objectives in a patient population representative of the entire patient population with GBM.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2017-10-31 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Mean ratio of detecting glioblastoma cancer between the Chaos Wand spectral readings and histopathology as ground truth | 6 months
  For participants newly diagnosed with glioblastoma multiforme or patients who are suspected of having glioblastoma on pre-operative imaging who consent to the use of the Chaos Wand during surgery, 15-20 spectral readings will be compared to histopathology as ground truth to measure the sensitivity of the Chaos Wand to detect glioblastoma. For example, if a patient has 15 spectral readings but only 13 are histologically consistent with cancer, then the sensitivity of the wand would be 13/15*100 = 87%. A mean value with standard deviation will be reported across all participants in the study.

SECONDARY OUTCOMES:
Number of participants experiencing post-operative intracranial hemorrhage following surgical resection of glioblastoma with use of the Chaos Wand during surgery | Up to 1 month following surgery
  For participants newly diagnosed with glioblastoma multiforme or are suspected of having glioblastoma based on pre-operative imaging who consent to the use of the Chaos Wand during surgery, the number of cases of intracranial hemorrhage during the post-operative hospital course will be measured.
Number of participants experiencing post-operative ischemic stroke following surgical resection of glioblastoma with use of the Chaos Wand during surgery | Up to 1 month following surgery
  For participants newly diagnosed with glioblastoma multiforme or are suspected of having glioblastoma based on pre-operative imaging who consent to the use of the Chaos Wand during surgery, the number of cases of ischemic stroke during the post-operative hospital course will be measured.
Number of participants experiencing post-operative surgical site infection following surgical resection of glioblastoma with use of the Chaos Wand during surgery | Up to 1 month following surgery
  For participants newly diagnosed with glioblastoma multiforme or are suspected of having glioblastoma based on pre-operative imaging who consent to the use of the Chaos Wand during surgery, the number of cases of surgical site infection during the post-operative hospital course will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Sughrue, MD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States